CLINICAL TRIAL: NCT06077591
Title: Prospective Clinical Validation of Next Generation Sequencing (NGS) and Patient-Derived Tumor Organoids (PDO) Guided Therapy in Patients with Advanced/ Inoperable Solid Tumors
Acronym: PDO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, MD, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prince of Wales Hospital
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention in this study is to perform tissue sampling to patient's tumor which are then subjected to DNA extraction for whole exome sequencing, organoid culture, and drug screen. This takes between 2- 4 weeks. In the interim period, the patient is allowed to receive a chemotherapy agent, a target agent or hormone therapy between the time of the biopsy and the availability of drug screen results. An MDT board will review the drug screen results and excluded drug choice of poor response. Then the referring oncologist has the final discretion on the choice of chemo- or targeted agent as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient-Derived Tumor Organoids (PDO) Guided Therapy (Experimental): Intervention in this study is to perform tissue sampling to patient's tumor which are then subjected to DNA extraction for whole exome sequencing, organoid culture, and drug screen. An MDT board will review the drug screen results and excluded drug choice of poor response. Then the referring oncologist has the final discretion on the choice of chemo- or targeted agent as usual.
  Interventions: Other: Patient-Derived Tumor Organoids

INTERVENTIONS:
Other: Patient-Derived Tumor Organoids — Intervention in this study is to perform tissue sampling to patient's tumor which are then subjected to DNA extraction for whole exome sequencing, organoid culture, and drug screen. An MDT board will review the drug screen results and excluded drug choice of poor response. Then the referring oncologist has the final discretion on the choice of chemo- or targeted agent as usual.

SUMMARY:
Precision oncology aims to improve clinical outcome of patients by offering personalized treatment through identifying druggable genomic aberrations within their tumors. This is particularly valid when it comes to offering alternative treatment options for patients with advanced tumors that are chemo-refractory. Patient-derived organoids (PDOs) are 3 dimensional tumoroids that can be expanded ex vivo and are both pheno- and genotypically identical to patients' tumors. Observational studies have shown that PDO-based drug screens can predict treatment response with high sensitivity and specificity. Vlachogiannis G. reported a living biobank of patient-derived organoids (PDOs) from patients with advanced GI cancers enrolled in clinical trials. PDOs can recapitulate patients' clinical response to chemotherapeutic agents. In 19 tumor organoids, the group performed molecular profiling and drug screens and then compared ex vivo organoid responses to anticancer drugs. Drug response to PDO based orthotopic mouse tumor xenografts correlated to the drug response of the patient in clinical trials. Further to the study, there were other retrospective validation studies utilizing PDOs from patients enrolled in clinical trials such as the TUMOROID, CinClare to predict clinical response. Ooft studied PDOs from patients with metastatic colorectal cancers enrolled in the TUMOROID study to predict response to irinotecan-based therapies. Yao generated a organoid biobank of 80 locally advanced rectal cancers. These patients were derived from a phase III study (CinClare) that compared neoadjuvant chemo-radiation using either capecitabine or CAPIRI. Response to chemoradiation in patients matched to that of rectal cancer organoids (sensitivity 78% and specificity 91.9%). In a systematic analysis of 17 studies (9 on advanced GI and pancreatic cancers, one on renal cell cancer and others on miscellaneous cancers), the pooled sensitivity and specificity for discriminating patients with a clinical response through PDO-based drug screen was 0.81 (95%CI 0.69-0.89) and 0.74 (95%CI 0.64-0.82) respectively. Within 4-6 weeks, PDO-based drug screen creates a true personalised platform by predicting patient-specific drug response with high accuracy. Recent technical advancements in growing these PDO 'avatars' from biopsies have made it possible to test suitable anticancer drugs in patients with advanced inoperable tumors, and explore the new possibilities for treatment options that otherwise would be missed by standard conventional therapies. In 2019, our group embarked on PDO research; investigators obtained tissues from patients with advanced/ inoperable solid tumors, and performing drug screens on these PDOs ex vivo. In several patients, investigators were able to identified drugs not otherwise used through sequencing data, and observed remarkable clinical response in patients with PDO responsive tumors. Investigators illustrate with cases that underwent PDO culture and drug screens. [ See appendix ] In the literature, the clinical utility of treatment based on PDO informed drug options has however not been fully established. Investigators therefore propose a phase 2 proof-of-concept clinical trial to evaluate efficacy of NGS/ PDO guided treatment in patients with inoperable or metastatic solid tumors..

DETAILED DESCRIPTION:
Under informed consents, patients undergo tissue sampling (radiologic, endoscopic or surgical excision). DNA is extracted from tissue and sent for whole-exome sequencing (WES), organoid culture and drug testing. DNA mutations in PDO models will be determined using whole-exome sequencing (WES). Mutational burden and driver genes profile will be assessed for similarities to those identified in primary cancers. The genetic data generated will be interpreted for response to FDA-approved molecular targeting drugs. Investigators would study PDO cultures resistant to available chemotherapeutic options. They would be of exceptional value to study sensitivity to targeted agents, providing alternative treatment options for chemo-refractory diseases. Based on past experience, project team has developed a Standard Operational Protocol (SOP) in the area and establish pipeline in integrative analysis with genome data. PDO Culture and Genome-guided Drug Screen.To ensure clinical usefulness of our platform, investigators aim to deliver drug options of each PDO within a meaningful timeframe. In this framework of typically 4-6 weeks, investigators shall generate organoids, study their molecular profile and undertake ex vivo drug screening that would allow us to individualize therapy for each patient. Eligible patients are seen in an MDT board where patients' case history, laboratory and radiologic results are reviewed. With informed consent to trial participation, the patient undergoes tissue sampling to his tumor (by radiologic, endoscopic, or surgical methods). Sampled tumors are then subjected to DNA extraction for whole exome sequencing, organoid culture, and drug screen. This takes between 2- 4 weeks. In the interim period, the patient is allowed to receive a chemotherapy agent, a target agent or hormone therapy between the time of the biopsy and the availability of drug screen results. An MDT will review the drug screen results and recommend the use of a drug with a response in a PDO. When several drugs are shown to be efficacious, the referring oncologist has the final discretion on the choice of chemo- or targeted agent.

Tumor assessments will be performed at baseline, every 8 weeks. Investigators report all adverse events and serious adverse events (SAE) based on the definitions in NCI CTCAE. Investigators report all SAEs to the Joint NTEC-CUHK CREC within 24 hours of their occurrence. Senior physicians at CREC adjudicated all SAEs.

Investigators aim to determine clinical efficacy of NGS/ PDO drug screen guided treatment in patients with inoperable/ advanced solid tumors refractory to conventional chemotherapy. Investigators correlate PDO drug response ex vivo to clinical response in these patients. Our hypothesis is that WES and PDO drug screen can accurately identify candidate drugs that will reduce tumor size and confer benefits in these patients.

Investigators assume a treatment response with standard treatment be around 10%. A PDO and NGS guided treatment will likely improve the response rate to about 30% or more. In the first stage, 10 patients will be accrued, If there is one or fewer response, in these 10 patients, the study will be stopped. Otherwise an additional 19 patients will be accrued for a total of 29. The null hypothesis will be rejected if 6 or more responses are observed in 29 patients. This design yields a type 1 error rate of 0.05 and a power of 80%. Investigators plan to enrol 40 or more patients over a period of 2 years, with the assumption that in about 20% of patients, PDO culture is unsuccessful.

ELIGIBILITY:
Inclusion Criteria:

* patients with metastatic, inoperable or advanced solid tumors who are refractory to at least one standard chemo- or targeted drugs.
* The disease is accessible for a biopsy (radiologic or endoscopic) or resection of a metastatic site.
* These patients are seen at a multidisciplinary tumor board meeting prior to referrals.
* aged >18 years, able to provide written consents to trial participation,
* with an Eastern cooperative oncology group performance status of 0 or 1,
* with measurable disease in accordance with response evaluation criteria in solid tumors (RECIST) version 1.1.
* deem suitable for standard chemo-therapy; i.e. with a normal neutrophil count, hemoglobin > 9g/dl, serum creatinine, <1.5 x upper limit of normal, bilirubin < 1.5 x normal, Aspartate and alanine aminotransferases (<3 x ULN or <5x
* those with liver metastasis) and with an ejection Fraction >50% of normal on echocardiography.

Exclusion Criteria:

* unable to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
tumor response | 6 months
  tumor response, partial or complete (>30% reduction in tumor size)

SECONDARY OUTCOMES:
rate of partial or complete response | 6 months
  rate of partial or complete response
rate of progression free survival survival | 6 months
  rate of progression free survival
rate of overall survival | 6 months
  rate of overall survival
success rate in PDO culture and drug screen | 6 months
  success rate in PDO culture and drug screen
rate of grade III/IV toxicities. | 6 months
  rate of grade III/IV toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: James Lau, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No
in progress

REFERENCES:
- [Background] van der Velden DL, Hoes LR, van der Wijngaart H, van Berge Henegouwen JM, van Werkhoven E, Roepman P, Schilsky RL, de Leng WWJ, Huitema ADR, Nuijen B, Nederlof PM, van Herpen CML, de Groot DJA, Devriese LA, Hoeben A, de Jonge MJA, Chalabi M, Smit EF, de Langen AJ, Mehra N, Labots M, Kapiteijn E, Sleijfer S, Cuppen E, Verheul HMW, Gelderblom H, Voest EE. The Drug Rediscovery protocol facilitates the expanded use of existing anticancer drugs. Nature. 2019 Oct;574(7776):127-131. doi: 10.1038/s41586-019-1600-x. Epub 2019 Sep 30. PMID 31570881
- [Background] Sato T, Stange DE, Ferrante M, Vries RG, Van Es JH, Van den Brink S, Van Houdt WJ, Pronk A, Van Gorp J, Siersema PD, Clevers H. Long-term expansion of epithelial organoids from human colon, adenoma, adenocarcinoma, and Barrett's epithelium. Gastroenterology. 2011 Nov;141(5):1762-72. doi: 10.1053/j.gastro.2011.07.050. Epub 2011 Sep 2. PMID 21889923
- [Background] van de Wetering M, Francies HE, Francis JM, Bounova G, Iorio F, Pronk A, van Houdt W, van Gorp J, Taylor-Weiner A, Kester L, McLaren-Douglas A, Blokker J, Jaksani S, Bartfeld S, Volckman R, van Sluis P, Li VS, Seepo S, Sekhar Pedamallu C, Cibulskis K, Carter SL, McKenna A, Lawrence MS, Lichtenstein L, Stewart C, Koster J, Versteeg R, van Oudenaarden A, Saez-Rodriguez J, Vries RG, Getz G, Wessels L, Stratton MR, McDermott U, Meyerson M, Garnett MJ, Clevers H. Prospective derivation of a living organoid biobank of colorectal cancer patients. Cell. 2015 May 7;161(4):933-45. doi: 10.1016/j.cell.2015.03.053. PMID 25957691
- [Background] . De Souza, N. Organoids. Nat. Methods 15, 23 (2018).
- [Background] Li M, Izpisua Belmonte JC. Organoids - Preclinical Models of Human Disease. N Engl J Med. 2019 Feb 7;380(6):569-579. doi: 10.1056/NEJMra1806175. No abstract available. PMID 30726695
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Background] Ooft SN, Weeber F, Dijkstra KK, McLean CM, Kaing S, van Werkhoven E, Schipper L, Hoes L, Vis DJ, van de Haar J, Prevoo W, Snaebjornsson P, van der Velden D, Klein M, Chalabi M, Boot H, van Leerdam M, Bloemendal HJ, Beerepoot LV, Wessels L, Cuppen E, Clevers H, Voest EE. Patient-derived organoids can predict response to chemotherapy in metastatic colorectal cancer patients. Sci Transl Med. 2019 Oct 9;11(513):eaay2574. doi: 10.1126/scitranslmed.aay2574. PMID 31597751
- [Background] Yao Y, Xu X, Yang L, Zhu J, Wan J, Shen L, Xia F, Fu G, Deng Y, Pan M, Guo Q, Gao X, Li Y, Rao X, Zhou Y, Liang L, Wang Y, Zhang J, Zhang H, Li G, Zhang L, Peng J, Cai S, Hu C, Gao J, Clevers H, Zhang Z, Hua G. Patient-Derived Organoids Predict Chemoradiation Responses of Locally Advanced Rectal Cancer. Cell Stem Cell. 2020 Jan 2;26(1):17-26.e6. doi: 10.1016/j.stem.2019.10.010. Epub 2019 Nov 21. PMID 31761724
- [Background] Wensink GE, Elias SG, Mullenders J, Koopman M, Boj SF, Kranenburg OW, Roodhart JML. Patient-derived organoids as a predictive biomarker for treatment response in cancer patients. NPJ Precis Oncol. 2021 Apr 12;5(1):30. doi: 10.1038/s41698-021-00168-1. PMID 33846504
- [Background] Loong HH, Wong AM, Chan DT, Cheung MS, Chow C, Ding X, Chan AK, Johnston PA, Lau JY, Poon WS, Wong N. Patient-derived tumor organoid predicts drugs response in glioblastoma: A step forward in personalized cancer therapy? J Clin Neurosci. 2020 Aug;78:400-402. doi: 10.1016/j.jocn.2020.04.107. Epub 2020 Apr 24. PMID 32340843
- [Background] Driehuis E, Kretzschmar K, Clevers H. Establishment of patient-derived cancer organoids for drug-screening applications. Nat Protoc. 2020 Oct;15(10):3380-3409. doi: 10.1038/s41596-020-0379-4. Epub 2020 Sep 14. PMID 32929210
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835